CLINICAL TRIAL: NCT04338191
Title: mFOLFOXIRI Versus mFOLFOX6 as Adjuvant Chemotherapy for Locally Advanced Colorectal Cancer Patients After Preoperative Treatment With Oxaliplatin (FANTASTIC): a Multicenter, Phase 3 Randomized Controlled Trial
Brief Title: mFOLFOXIRI Versus mFOLFOX6 as Adjuvant Chemotherapy for Locally Advanced Colorectal Cancer
Acronym: FANTASTIC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIHSYSU-19
Record Dates: First submitted 2020-04-05; First posted 2020-04-08 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Colorectal Cancer
Keywords: Adjuvant chemotherpay; FOLFOXIRI
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Irinotecan; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mFOLFOXIRI adjuvant chemotherapy (Experimental): Patients will receive mFOLFOXIRI once every two weeks for 6 cycles as adjuvant chemotherapy
  Interventions: Drug: mFOLFOXIRI adjuvant chemotherapy
- mFOLFOX6 adjuvant chemotherapy (Active Comparator): Patients will receive mFOLFOX6 once every two weeks for 6 cycles as adjuvant chemotherapy
  Interventions: Drug: mFOLFOX6 adjuvant chemotherapy

INTERVENTIONS:
Drug: mFOLFOXIRI adjuvant chemotherapy — mFOLFOXIRI (oxaliplatin 85 mg/m2, irinotecan 150 mg/m2, and folinic acid 400 mg/m2 followed by 5-fluorouracil 2400mg/m2 as a 46-hour continuous infusion on day 1) for 6 cycles
  Other Names: Oxaliplatin; Irinotecan; Leucovorin; 5-Fluorouracil
  Arms: mFOLFOXIRI adjuvant chemotherapy
Drug: mFOLFOX6 adjuvant chemotherapy — mFOLFOXIRI (oxaliplatin 85 mg/m2, and folinic acid 400 mg/m2 followed by 5-fluorouracil 400mg/m2 infusion, and 2400mg/m2 as a 46-hour continuous infusion on day 1) for 6 cycles
  Other Names: Oxaliplatin; Leucovorin; 5-Fluorouracil
  Arms: mFOLFOX6 adjuvant chemotherapy

SUMMARY:
The current standard treatment for locally advanced rectal cancer is still fluorouracil-based neoadjuvant radiotherapy and chemotherapy followed by TME surgery, followed by adjuvant chemotherapy. Fluorouracil single-agent simultaneous sensitization of radiotherapy and chemotherapy has a pCR of about 15-20% and a tumor downgrade (ypStage 0-I) rate of about 35%. However, about 30% of patients still have distant metastasis, which is the main obstacle affecting the survival prognosis of patients with locally advanced rectal cancer.

About 50% -65% of patients was still stage II-III after neoadjuvant therapy. The long-term follow-up shows that for patients with ypT4 after surgery, the 3-year DFS is about 50%. For patients with ypN2, the 3-year DFS is less than 40%. Therefore, it is necessary to strengthen postoperative adjuvant chemotherapy to improve the survival prognosis for these patients.

Although FOLFOX adjuvant chemotherapy improved survival benefit than 5FU as adjuvant treatment in ypStage II-III patients after neoadjuvant treatment in ADORE trial. However, with the progress of neoadjuvant therapy research, more and more studies have proposed to move part or all of postoperative adjuvant chemotherapy to preoperative neoadjuvant therapy due to low compliance of adjuvant chemotherapy.

During neoadjuvant treatment, induction chemotherapy with FOLFOX / CAPEOX or consolidation therapy after CRT with FOLFOX / CAPEOX had been investigated a lot. The pCR rate was 19% -38%, and the tumor downstaging rate was about 50%. Another 50% of patients still had ypstage II-III postoperatively. The 3-year DFS for ypStage III was only 55% even with FOLFOX as adjuvant chemotherapy. And for ypT4N0 patients with ypstage IIB-IIC, there is also a higher risk of recurrence and metastasis. And it is urgent to explore new treatment strategies to improve this part of patients Survival prognosis.

For locally advanced colon cancer, surgery combined with postoperative adjuvant chemotherapy is currently the standard treatment mode for stage II-III colon cancer. About 30% of patients with locally advanced disease will relapse within 3 years, of which distant metastases are more common and eventually become the main cause of death of patients. For locally advanced colon cancer with a preoperative staging of T4b, the NCCN guidelines recommend surgery after neoadjuvant chemotherapy with FOLFOX or CAPOX regimens. In the FOxTROT study of neoadjuvant treatment of locally advanced colon cancer, for patients with T3> 5mm or T4, after 4 courses of neoadjuvant chemotherapy with FOLFOX regimen, 20.5% of patients still have T4 after surgery, and 15.2% of patients had N2 disease. For this part of patients, new postoperative treatment options should also be explored to improve patient survival and prognosis.

In view of the high efficiency of the three-agent FOLFOXIRI regimen in advanced colorectal cancer and the success in adjuvant chemotherapy after pancreatic cancer surgery, 5FU, oxaliplatin combined with irinotecan may have a synergistic effect. At present, a phase III randomized controlled study (IROCAS study) in Europe is underway. For high-risk phase III patients, the mFOLFOXIRI regimen is compared with mFOLFOX6 regimen adjuvant chemotherapy.

Based on the above reasons, our center plans to further carry out "multi-center, randomized, controlled phase III clinical study of mFOLFOXIRI versus mFOLFOX6 adjuvant chemotherapy after neoadjuvant oxaliplatin in locally advanced colorectal cancer." Improve the survival prognosis of postoperative high-risk colorectal cancer patients after neoadjuvant therapy.

DETAILED DESCRIPTION:
This trial is a two-arm, multicenter, open labelled, prospective, randomized phase III studies. Eligible patients with locally advnaced colorectal cancer receiving oxlipaltin-based (less than 3 months) noeadjuvant treatment, the postoperative stage was high-risk stage II (ypT4N0M0) or stage III (ypTanyN1-2M0). These high risk patients will be randomly assigned, in a 1:1 ratio, to receive either mFOLFOXIRI or FOLFOX for 3 months as adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* ECOG PS 0-1
* Exposure to Oxaliplatin in preoperative treatment (less than 3 months)
* Induction or consolidation chemotherapy in rectal cancer or Concurrent FOLFOX with CRT in rectal cancer
* Neoadjuvant treatment with CAPOX or FOLFOX in colon cancer
* Curative surgery (R0 resection)
* ypStage IIB, IIC and ypStage III
* No distant metastasis after surgery
* ≤ 8 weeks prior to randomization

Exclusion Criteria:

* Previous or concurrent cancer that is distinct in primary site or histology from colon cancer within 5 years prior to randomization.
* Significant cardiovascular disease including unstable angina or myocardial infarction within 6 months before initiating study treatment.
* Heart failure grade III/IV (NYHA-classification).
* Unresolved toxicity higher than CTCAE v.4.0 Grade 1 attributed to any prior therapy/procedure.
* Subjects with known allergy to the study drugs or to any of its excipients.
* Current or recent (within 4 weeks prior to starting study treatment) treatment of another investigational drug or participation in another investigational study.
* Breast- feeding or pregnant women
* Lack of effective contraception

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 638 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
3-year Disease-free survival | up to 3 years
  Defined as the time from randomization to relapse or death, whichever occurred first

SECONDARY OUTCOMES:
Overall survival | up to 5 years
  Defined as the time from randomization to death from any cause
The grade of toxicity will be assessed using the NCI common toxicity criteria, version 5.0. | up to 3 years
  Safety
QLQ-C30 Quality of Life questionnaire | up to 3 years
Quality of Life assessed by SF-36 | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Yanhong Deng, Ph.D, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Gastrointestinal Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China